CLINICAL TRIAL: NCT06145555
Title: Acute Psychological Sleep Stabilisation for Patients Hospitalised With Depression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Sandra Tamm, M.D., PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2023-02223-01
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Insomnia; Depression
Keywords: CBT; Psychiatry; Inpatient care; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute psychological sleep stabilization (Experimental): The basis of the treatment is CBT-I adapted to a short version performed by trained staff (nurses or mental health care assistants) together with a psychologist. The manuals are designed to be read by patients and staff together and each treatment manual covers a specific topic. The focus of the treatment is behavioral changes and central manuals are stimulus control and scheduled sleep and sleep compression (if needed).
  Interventions: Behavioral: Acute psychological sleep stabilization
- Sleep hygiene education (Active Comparator): The control treatment is delivered through structured manuals which patients work through together with the staff. The manuals cover sleep hindering factors (eg coffee, nicotine), sleep promoting factors (eg physical activity during the day, relaxation, blinds), sleep aids (for example, weight blanket, calm music).
  Interventions: Behavioral: Sleep hygiene education

INTERVENTIONS:
Behavioral: Acute psychological sleep stabilization — See above (arm description)
  Arms: Acute psychological sleep stabilization
Behavioral: Sleep hygiene education — See above (arm description)
  Arms: Sleep hygiene education

SUMMARY:
Disturbed sleep occurs in almost all patients in psychiatric inpatient care, and although it is well known that comorbid sleep disorders in depression often persist after treatment of depression and also increase the risk of new depressive episodes, the availability of effective, evidence-based treatments for sleep disorders in hospitalised patients is very limited.

The overall goal of the current project is to translate, adapt and evaluate an acute psychological sleep treatment based on cognitive behavioural therapy for insomnia (CBT-I) for patients hospitalized with depression and comorbid sleep problems in the specialized psychiatric inpatient care in the Stockholm Region. The main hypothesis for the study is that acute psychological sleep stabilization (APS) reduces self-reported sleep complains compared to care as usual reinforced with sleep hygiene advice, and secondary hypotheses are that APS also leads to reduced depressive symptoms and earlier discharge.

The project includes a pilot study, which will be followed by a randomized, controlled trial of APS compared to care as usual with structured sleep hygiene (minimal active control) and treatment effect is evaluated every three days during the hospital stay and 1,2,4 and 12 weeks after randomization. APS will be performed by existing staff in the department with the support of a psychologist.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the psychiatric inpatient care (Psykiatri Sydväst)
* Depressive symptoms / confirmed depressive episode (uni- or bipolar)
* Reports or is observed to have sleep problems in the form of insomnia, hypersomnia or delayed circadian phase
* Knowledge of Swedish or English that is deemed sufficient to undergo the treatment
* Consent to be included in the study and is judged to have understood what the study entails (care according to the Compulsory Psychiatric Care Act is not in itself an exclusion criterion)

Exclusion Criteria:

* Dementia
* Intellectual disability
* Severe somatic comorbidity with life expectancy <6 months
* Ongoing mania / mixed-state
* Complex problems that make APS impossible or inappropriate
* Expected discharge within 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | 2 weeks post randomization (secondary timepoints include day 4, 7, 10 and week 4 and 12)
  A self-report measure of insomnia symptoms. 7-item, self-rated questionnaire measuring insomnia severity. Total score 0-28, higher score indicates more severe sleep problems.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Day 4, 7, 10 14 and week 4 and 12 post randomisation
  Self-reported depressive symptoms. PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. Total score 0-27, higher score indicates more severe depressive symptoms.
Generalised Anxiety Disorder 7-item scale (GAD-7) | Day 4, 7, 10 14 and week 4 and 12 post randomisation
  Self-reported anxiety symptoms. A seven-item instrument that is used to measure or assess the severity of generalised anxiety disorder/symptoms. Total score 0-27. Higher scores indicative of more severe problem.
European Quality of Life 5 Dimensions scale (EQ-5D) | Week 2, 4 and 12 post randomisation
  Self-reported quality of life. An instrument which evaluates the generic quality of life developed in Europe and widely used. The scale comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.

OTHER OUTCOMES:
Sleep Diary | 0-14 days post randomisation
  Participants will report their bedtime, risetime, amount of sleep daily using a simplified version of a sleep diary. We will look at total sleep time, sleep efficiency, and timing of sleep.
Actigraphy | 0-14 days post randomisation
  An actigraph is placed on the participant's arm for 2 weeks. It measures participants' arm-movements. An algorithm can be used to estimate sleep from movement data.Data from actigraphs will be reported and analysed
Side effects of treatment | Day 7 and 14 post randomisation
  Patients will be asked to report any side-effects of the treatment with an open question
Treatment Credibility Scale | Day 4 post randomisation
  A five-item version of Credibility/Expectancy Questionnaire, total score ranging from 0-50. Higher scores indicative of higher credibility.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Tamm, Principal Investigator — Karolinska Institutet; Susanna Jernelöv, Principal Investigator — Karolinska Institutet
Locations (1):
- Psykiatri Sydväst, Karolinska Hospital Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared